CLINICAL TRIAL: NCT05016388
Title: Evaluation of the Efficacy of a Multidimensional Collaborative Model to Improve the Resolution of Depression in Primary Care Teams in the Maule Region
Brief Title: Collaborative Multidimensional Intervention for Depression in Chile
Acronym: CMID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Talca (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA20I0031
Record Dates: First submitted 2021-07-30; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-06

CONDITIONS: Depression
Keywords: Complex Depression; Collaborative Model; Primary Health Care; Trauma Informed Care; Difficult to treat Depression
MeSH Terms: conditions — Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The collaborative multidimensional model (CMD) for depression incorporates to the current knowledge for the treatment of depression in primary care (PHC) teams in Chile, competences for the management of clinical, functional, psycho-biographical dimensions. These dimensions are prevalent in patients consulting PHC in Chile, associated to a complex depression sub-type, for which the current clinical guide does not provide recommendations. The implementation of this model entails a 22-hour training consisting of lectures and workshops through a virtual platform, followed by the application of the CMD in the PHC teams. In brief, the application of the model involves the creation of a case manager that prioritizes participants according to their complexity and collaboration sessions with the participation of specialists and the PHC team every 15 days for at least 3 months after the training.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Principal Investigator will not receive information about the assigned group (intervention/control). The Outcome assessor will be blinded to the assigned group (intervention/control) for data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Multidimensional Model (CMD) (Experimental): The teams in the CMD group will be composed each of at least a MD, a psychologist, and a social worker. The teams will receive the CMD training and the CMD will be installed in the primary health care (PHC) center. Then, the participants with depression who enter treatment for depression in their respective PHC center, will be enrolled and evaluated by an external team, blind to the interventions at the beginning, three and six months after.
  Interventions: Other: Collaborative Multidimensional Model (CMD)
- Standard Model (SM) (Other): The teams in the SM group will be composed each of at least a MD, a psychologist, and a social worker. The teams will receive the SM training and the SM will be set in the primary health care (PHC) center. Then, the participants with depression who enter treatment for depression in their respective PHC center, will be enrolled and evaluated by an external team, blind to the interventions at the beginning, three and six months after.
  Interventions: Other: Standard Model (SM)

INTERVENTIONS:
Other: Collaborative Multidimensional Model (CMD) — The teams enrolled in the CMD intervention will have a 22-hour training that integrates current knowledge of depression with skills for the management of functional variables, interpersonal, social, emotional regulation, and history of biographical adversity from childhood considering the trauma informed care paradigm. After the training, the PHC teams will implement the depression treatment according to a collaborative model.
  Other Names: Intervention
  Arms: Collaborative Multidimensional Model (CMD)
Other: Standard Model (SM) — The teams enrolled in the SM intervention will have a 22-hour training that integrates the current national clinical guide for Depression in Chile. This guide offers a staggered treatment according to the severity of the depression. After the training, the PHC teams will implement the depression treatment according to the SM.
  Other Names: Control
  Arms: Standard Model (SM)

SUMMARY:
This study protocol aims to determine the efficacy of a collaborative multidimensional model (CMD) to improve the results of depression in primary care (PHC) in Chile. The CMD includes training of PHC teams, on the recognition of clinical, functional and psycho-biographic dimensions associated to a complex depression sub-type, difficult to treat, prevalent in PHC in Chile, for which there are no recommendations in current clinical guidelines. This model implies the implementation of a collaborative model, trauma informed care, patient- centered, that includes a case manager, the use of instruments and a close relationship between the PHC team and the specialty level. At least twelve primary care teams belonging to the Maule Region will be randomly assigned to one of the two arms of the study, the CMD group and the current standard model (SM). After the implementation of the CMD, an intentional sample of 394 participants who agreed to participate, with prior informed consent, will be evaluated by a blind research team at the beginning, at three and six months with a battery of instruments. An improvement in depressive symptoms, anxiety and functional variables is expected in participants treated in CMD versus SM. This protocol was approved by the Research Ethics Council of the University of Talca, Talca. The goal is to publish the preliminary results in December 2022.

DETAILED DESCRIPTION:
The research design is a cluster randomized clinical trial. Inter-professional teams from at least 12 primary care centers of the Maule area will be randomized in two arms: intervention and control. The intervention arm will receive a training in the collaborative multidimensional model for depression (CMD) and the control arm will be trained in the current clinical guide (SM).

After the CMD implementation, a sample of 394 participants entered to treatment for depression at their respective center will be invited to participate. This sample has been calculated estimating a maximum error of 5 %, a confidence level of 95 %, a power of 80 % a maximum variance of 50 % and a retention of 85 %.

The patients who agreed to participate, will be treated by their respective PHC team and their therapeutic indications will be included in the official clinical records for each participant. Also these patients, after informed consent, will be evaluated by a blind external research team at the beginning, at three and six months with a battery of instrument.

The informed consents will be kept in locked folders. The data obtained by the external evaluators will be confidential, entered into a virtual spreadsheet in a coded form on a server of the U. of Talca through a personal computer. Participant's diagnoses will be coded using the MINI.

A protocol for the management of adverse situations of an emergency nature will be provided.

The results will be presented according to the CONSORT guide for randomized clinical trials, with its extensions to cluster and non-pharmacological interventions.

Analysis of the primary and secondary outcomes will be performed by intention to treat. In the initial analysis, the balance between the characteristics of the different samples will be evaluated and a linear multi-variable regression will be performed to establish differences at 3 and 6 months, adjusting the results according to the initial data, in case of imbalance for all outcomes. A sensitivity analysis based on different assumptions will also be implemented, to investigate the possible effects of missing data. Statistical analysis will be done with SPSS software.

The research protocol was approved by the Ethics Committee of the University of Talca and approved by the Agencia Nacional de Investigación y Desarrollo (ANID), the national institution that audit the project through a follow-up sheet and yearly controls.

ELIGIBILITY:
Inclusion Criteria:

* Starting the treatment for depression in Primary Care according the Health Guarantees.
* Confirmed depression diagnosis according to the Mini International Diagnostic Interview Mini International Neuropsychiatric Interview (MINI, Sheehan et al. 1998).

Exclusion Criteria:

* Sensory disability
* Inability to provide the informed consent
* not having contact phone number
* Continuing treatment for depression
* High suicidal risk
* Suspected bipolar and psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive symptoms at three months relative to baseline | Three months after admission to depression treatment
  Depressive symptoms will be assessed by the Patient Health Questionnaire (PhQ9).
  The Patient Health Questionnaire is a nine-item self-report measure that assesses the presence of depressive symptoms based on the DSM-IV criteria for major depressive. The Spanish version of the Patient Health Questionnaire has been validated in Chile.
  The Patient Health Questionnaire measures the symptoms experienced by the patients during the two weeks prior to the interview.
  Total score ranges from 0 to 27 points and greater scores means worse symptoms.
Change in Depressive symptoms at six months relative to baseline | Six months after admission to depression treatment
  Depressive symptoms will be assessed by the Patient Health Questionnaire (PhQ9).
  The Patient Health Questionnaire is a nine-item self-report measure that assesses the presence of depressive symptoms based on the DSM-IV criteria for major depressive. The Spanish version of the Patient Health Questionnaire has been validated in Chile.
  The Patient Health Questionnaire measures the symptoms experienced by the patients during the two weeks prior to the interview.
  Total score ranges from 0 to 27 points and greater scores means worse symptoms.

SECONDARY OUTCOMES:
Change in Anxiety symptoms at three months relative to baseline | Three months after admission to depression treatment
  Anxiety symptoms will be evaluated by the generalized anxiety scale-7 (GAD/7 validated in Spanish).
  The generalized anxiety scale-7 serve as screening for generalized anxiety disorder.
  The generalized anxiety scale-7 is a 7 Likert-type items with response options from 0 to 3 points .
  A total score ranges from 0 to 21 points, greater scores means worse anxiety symptoms.
Change in Anxiety symptoms at six months relative to baseline | Six months after admission to depression treatment
  Anxiety symptoms will be evaluated by the generalized anxiety scale-7 (GAD/7 validated in Spanish).
  The generalized anxiety scale-7 serve as screening for generalized anxiety disorder.
  The generalized anxiety scale-7 is a 7 Likert-type items with response options from 0 to 3 points .
  A total score ranges from 0 to 21 points, greater scores means worse anxiety symptoms.
Change in Interpersonal Dysfunction and Social Dysfunction at three months relative to baseline | Three months after admission to depression treatment
  Interpersonal and social areas will be evaluated by the sub-scales of the Outcome Questionnaire (OQ-45) interpersonal and social role.
  The Outcome Questionnaire version 45-2 (OQ-45) is a self-administered instrument with evaluations in interpersonal and social role with Lkert-items whose response options range from 0 to 4 points.
  The interpersonal subscale includes 12 items with scores that range from 0 to 48 points and the social scale includes 9 items with scores that range from 0 to 36 points. Greater score means worse Interpersonal and social function.
Change in Interpersonal Dysfunction and Social Dysfunction at six months relative to baseline | Six months after admission to depression treatment
  Interpersonal and social areas will be evaluated by the sub-scales of the Outcome Questionnaire (OQ-45) interpersonal and social role.
  The Outcome Questionnaire version 45-2 (OQ-45) is a self-administered instrument with evaluations in interpersonal and social role with Likert-items whose response options range from 0 to 4 points.
  The interpersonal subscale includes 12 items with scores that range from 0 to 48 points and the social scale includes 9 items with scores that range from 0 to 36 points. Greater score means worse Interpersonal and social function.
Change in Emotion Regulation at three months relative to baseline | Three months after admission to depression treatment
  Difficulties in Emotion regulation will be evaluated by the Emotion Regulation Scale (ERS) validated in Chile.
  The Emotion Regulation Scale assesses emotions with respect to control, rejection, inattention, interference, and confusion.
  ERS scale consists of 28 items with a Likert-type response options from 1 to 5 points, the scores range from 0 to 140 points and greater scores indicate worse emotional regulation.
Change in Emotion Regulation at six months relative to baseline | Six months after admission to depression treatment
  Difficulties in Emotion regulation will be evaluated by the Emotion Regulation Scale (ERS) validated in Chile.
  The Emotion Regulation Scale assesses emotions with respect to control, rejection, inattention, interference, and confusion.
  ERS scale consists of 28 items with a Likert-type response options from 1 to 5 points, the scores range from 0 to 140 points and greater scores indicate worse emotional regulation.
Therapeutic adherence at three months | Three months after admission to depression treatment
  Adherence to treatment will be evaluated by the Scale of Adherence to General Health Treatment validated in Chile.
  The scale of Adherence consists of 21 questions with a Likert scale whose response options range from 1 to 6 points adding up to a total score from 22 to 132, lesser score means worst therapeutic adherence.
Therapeutic adherence at six months | Six months after admission to depression treatment
  Adherence to treatment will be evaluated by the Scale of Adherence to General Health Treatment validated in Chile.
  The Scale of Adherence consists of 21 questions with a Likert scale whose response options range from 1 to 6 points adding up to a total score from 22 to 132, lesser score means worst therapeutic adherence.

OTHER OUTCOMES:
Self-efficacy of the primary care mental health team at baseline | Baseline (at the first training session)
  The self-efficacy of the primary care mental health team will be evaluated by the general self-efficacy scale (GSES) validated in Chile.
  The general self-efficacy scale consists of a 10-item Likert scale with response options from 1 to 7 points.
  To total score ranges from 1 to 70 points with greater scores meaning greater self efficacy.
Self-efficacy of the primary care mental health team after three months | Three months after the first training session
  The self-efficacy of the primary care mental health team will be evaluated by the general self-efficacy scale (GSES) validated in Chile.
  The general self-efficacy scale consists of a 10-item Likert scale with response options from 1 to 7 points.
  To total score ranges from 1 to 70 points with greater scores meaning greater self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica G Vitriol, MD, Study Director — University of Talca; Alfredo A Cancino, MD, Study Director — University of Talca; Maria L Aylwin, PhD, Principal Investigator — University of Talca

IPD SHARING:
Plan to Share IPD: Yes
The sharing of the IPD data requires the authorization of the Ethics committee of the Universidad de Talca.
  The Study protocol, Statistical Analysis Plan, Informed Consent, Clinical Study Report and Analytic code will be included in future publications.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From September 2022 to March 2023 the data will be available through web platforms like Mendely Data
Access Criteria: The data published will be shared through web platforms like Mendely Data and further data may be shared by special request to the principal researcher

REFERENCES:
- [Background] Saldivia S, Aslan J, Cova F, Vicente B, Inostroza C, Rincon P. [Psychometric characteristics of the Patient Health Questionnaire (PHQ-9)]. Rev Med Chil. 2019;147(1):53-60. doi: 10.4067/S0034-98872019000100053. Spanish. PMID 30848765
- [Background] Clavijo M, Yevenes F, Gallardo I, Contreras AM, Santos C. [The general self-efficacy scale (GSES): Reevaluation of its reliability and validity evidence in Chile]. Rev Med Chil. 2020 Oct;148(10):1452-1460. doi: 10.4067/S0034-98872020001001452. Spanish. PMID 33844715
- [Background] von Bergen, A., & de la Parra, G. (2002). OQ-45.2, Cuestionario para evaluación de resultados y evolución en psicoterapia: Adaptación, validación e indicaciones para su aplicación e interpretación [OQ-45.2, An Outcome Questionnaire for Monitoring Change In Psychotherapy: Adaptation, Validation and Indications for its Application and Interpretation]. Terapia Psicológica, 20(2), 161-176.
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Guzman-Gonzalez M, Mendoza-Llanos R, Garrido-Rojas L, Barrientos J, Urzua A. [Cut-off points of the difficulties in Emotion Regulation Scale for the Chilean population]. Rev Med Chil. 2020 May;148(5):644-652. doi: 10.4067/S0034-98872020000500644. Spanish. PMID 33399757
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] McAllister-Williams RH, Arango C, Blier P, Demyttenaere K, Falkai P, Gorwood P, Hopwood M, Javed A, Kasper S, Malhi GS, Soares JC, Vieta E, Young AH, Papadopoulos A, Rush AJ. The identification, assessment and management of difficult-to-treat depression: An international consensus statement. J Affect Disord. 2020 Apr 15;267:264-282. doi: 10.1016/j.jad.2020.02.023. Epub 2020 Feb 7. PMID 32217227
- [Background] Archer J, Bower P, Gilbody S, Lovell K, Richards D, Gask L, Dickens C, Coventry P. Collaborative care for depression and anxiety problems. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD006525. doi: 10.1002/14651858.CD006525.pub2. PMID 23076925
- [Background] Raja S, Hasnain M, Hoersch M, Gove-Yin S, Rajagopalan C. Trauma informed care in medicine: current knowledge and future research directions. Fam Community Health. 2015 Jul-Sep;38(3):216-26. doi: 10.1097/FCH.0000000000000071. PMID 26017000
- [Background] Vitriol V, Cancino A, Serrano C, Ballesteros S, Potthoff S. Remission in Depression and Associated Factors at Different Assessment Times in Primary Care in Chile. Clin Pract Epidemiol Ment Health. 2018 Mar 26;14:78-88. doi: 10.2174/1745017901814010078. eCollection 2018. PMID 29643931
- [Background] Vitriol V, Cancino A, Serrano C, Ballesteros S, Ormazabal M, Leiva-Bianchi M, Salgado C, Caceres C, Potthoff S, Orellana F, Asenjo A. Latent Class Analysis in Depression, Including Clinical and Functional Variables: Evidence of a Complex Depressive Subtype in Primary Care in Chile. Depress Res Treat. 2021 Feb 11;2021:6629403. doi: 10.1155/2021/6629403. eCollection 2021. PMID 33628499
- [Background] Salvo G L. [Magnitude, impact and recommended management strategies for depression, with reference to Chile]. Rev Med Chil. 2014 Sep;142(9):1157-64. doi: 10.4067/S0034-98872014000900010. Spanish. PMID 25517056
- [Derived] Vitriol V, Cancino A, Sciolla A, Guinez S, Calvo J, Ormazabal M, Kreither J, Ballesteros S, Aylwin ML. Effectiveness of a multidimensional collaborative approach versus usual care in the treatment of adult depression in primary care in Chile: study protocol for a single blinded cluster randomized controlled trial. F1000Res. 2024 Oct 11;11:203. doi: 10.12688/f1000research.75764.2. eCollection 2022. PMID 39464248